CLINICAL TRIAL: NCT03857802
Title: Efficiency of a Nursing Intervention in Sleep Hygiene in Prediabetes and Diabetes Mellitus 2
Brief Title: Efficiency of a Nursing Intervention in Sleep Hygiene
Acronym: ENISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Cristina García Serrano, Nurse of Primary Care, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JordiGol
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-01

CONDITIONS: Sleep Disorder; Metabolic Glucose Disorders
Keywords: diabetes mellitus type 2; prediabetic state; sleep hygiene; haemoglobin A glycosylated; clinical nursing research
MeSH Terms: conditions — Sleep Wake Disorders; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Prediabetic State; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Experimental study, non-masked clinical trial of evaluation of an educational intervention in the field of Primary Care Nursing: Basic Health Area (BHA) of Balaguer. Two groups will be established randomly: experimental group and control group. In the experimental group will proceed to the explanation of sleep hygiene measures to improve the quality of sleep. In the control group, the same follow-up visits and the same blood extractions will be carried out, but no educational activity on sleep will be carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep hygiene intervention (Experimental): In the experimental group will proceed to the explanation of sleep hygiene measures to improve the quality of sleep. After 3 months, at the next health check, the quality of sleep questionnaire will be carried out together with the blood extraction.
  Interventions: Behavioral: Sleep hygiene intervention
- No sleep hygiene intervention (No Intervention): In the no intervention group, the same follow-up visits and the same blood extractions will be carried out, but no educational activity on sleep will be carried out.

INTERVENTIONS:
Behavioral: Sleep hygiene intervention — An individual education will be carried out following a bidirectional feedback method. It is intended to develop skills to make conscious and autonomous decisions. The explanation will consist:
  1. Information and reading with discussion of the educational sheet: The 9 tips for a healthy sleep will be read, point by point. The nurse will be open to discuss those that generate doubt.
  2. Confrontation: even if the patient does not ask any questions about it, it will be necessary to ask if he has understood the advice.
  3. Participated information: Questions will be asked to the patient such as: "Did you already know any of these tips?".
  A telephone call per month will be made as an educational reinforcement to the intervention.
  Arms: Sleep hygiene intervention

SUMMARY:
Background: The relationship between the appearance of insulin resistance phenomena and insufficient or poor-quality sleep is scientifically documented.

Objectives: To determine the effectiveness of an intervention based on behavioural techniques on sleep in the nursing consultation in the Primary Care setting to improve the level of HbA1c in patients diagnosed with diabetes mellitus 2 (DM2) or prediabetes.

Hypothesis: Patients diagnosed with DM2 or prediabetes with poor sleep quality would improve their HbA1c levels after an intervention on healthier sleep hygiene practices. Sleeping 6 or less hours in adults diagnosed with DM2 or prediabetes would be related to worse metabolic control results. Patients diagnosed with DM2 or prediabetes who would value their sleep as poor quality would have poorer metabolic control.

Methodology: Design: Not masked randomized clinical trial. Target population: Patients diagnosed up to the time of DM2 (E11) or prediabetes (R73, R73.9) with age over 18 attending the chronic nurses' follow-up visits of the Basic Health Area of Balaguer in the time range from November 2017 to December 2018. Determinations: Dependent variables: Glycemia and HbA1c. Independent variables: Sex, age, value of the Pittsburgh Sleep Quality Index (PSQI), declared hours of sleep, sleep efficiency, body mass index (BMI), pharmacologic antidiabetic treatment, changes in it, changes in diet, physical exercise and sleep hygiene. Statistical analysis: Analysis of the comparability of the groups and calculation of the confidence interval of the difference in the glycaemic values and HbA1c at the end of the follow-up, with respect to the initiation within the intervention group and within the control, and control group with respect to the group intervention.

DETAILED DESCRIPTION:
Several studies have shown the association between short and poor sleep quality and alterations in glucose metabolism as well as the appearance of insulin resistance phenomena. This issue makes the research on this subject relevant to establish interventions aimed at improving the quality of sleep. Nursing professionals in the field of Primary Care have a decisive role in the monitoring and control of chronic diseases, among which DM2 stands out due to its high prevalence, great morbidity and mortality and healthcare pressure. Therefore, it is necessary to check the efficiency of healthy sleep hygiene to carry out prevention and achieve good metabolic control of the patient. Therefore, it is, in this way, important to prevent the development of the disease in the case of patients with prediabetes and the appearance of complications in patients with DM2.

Therefore, the overall objective is to determine the efficiency of an intervention based on behavioural techniques on sleep in the nursing consultation in the Primary Care setting to improve the level of HbA1c in patients diagnosed with DM2 or prediabetes.

The specific objectives are:

1. Describe the mean and range of hours that patients with DM2 or prediabetes declare to sleep.
2. To analyse the assessment of the quality of sleep referred by people with DM2 or prediabetes through the PSQI.
3. Calculate the correlation between the number of hours of sleep declared and the HbA1c values.
4. Compare the amount and quality of sleep and HbA1c value in the control group and the experimental group.

   In the other hand, the hypotesis are:

   -Patients diagnosed with DM2 or prediabetes with poor sleep quality would improve their HbA1c levels after an intervention on healthier sleep hygiene practices.
   * Sleeping 6 or less hours in adults diagnosed with DM2 or prediabetes would be related to worse results of metabolic control.
   * Patients diagnosed with DM2 or prediabetes who would value their sleep as poor quality would have worse metabolic control.

   The variables are:

   Dependent variable:
   * Value of the difference between the basal glycemia figure at the beginning and at the end of the study. Measurement in mg / dL.
   * Value of the difference between the HbA1c level at the beginning and at the end of the study. Measure in%.

   Independent variable:
   * Age. Measure in years.
   * Sex. Man/Woman.
   * Diagnosis (International Classification of Diseases, 10th version). E11 Non-insulin-dependent Diabetes Mellitus/R73 Elevated blood glucose level/ R73.9 Hyperglycaemia, unspecified.
   * Antidiabetic pharmacological treatment. Yes/No.
   * BMI. Measure in kg/m2. PSQI (pre and post-intervention). Good sleep quality (≤ 5 points)/ Bad sleep quality (> 5 points).
   * Declared sleeping hours (pre and post-intervention). Measure in hours/day.
   * Sleeping efficiency (pre and post-intervention). Measure in%
   * Change in antidiabetic pharmacological treatment 3 months after the first visit. Yes/No
   * Change in diet 3 months after the first visit. Yes/No.
   * Change in physical exercise 3 months after the first visit. Yes/No.
   * Change in sleep hygiene (post-intervention). Yes/No.

   The data will be collected through the computerized clinical record ECAP and through the patient's own consent and acceptance of their participation in the study.

   Necessary data for the selection of the sample:

   - Computerized clinical and administrative database (ECAP) of the participating centres: this source will be used to obtain the complete list of patients with the diagnostic codes E11 (E11.2-E11.9), R73 and R73.9 and the criterion of age (≥ 18 years).

   Necessary data to obtain the values of the dependent variables:

   - HbA1c and baseline glycaemia values for the experimental group and control group performed pre and post-intervention. The results of the analytics will be obtained, according to laboratory criteria.

   Necessary data to obtain the values of the independent variables:
   * Declared sleep hours, efficiency and quality of sleep from the PSQI performed on the patient. The average number of hours of sleep on weekdays will be requested at the time of introducing the individual into the study regardless of whether the individual is active or a pensioner. The values will be recorded in the initial and final visit through the PSQI.
   * BMI obtained in the nursing consultation in the follow-up visits before 6 months from the date of the visit. Otherwise, it will be calculated after the measurement of weight and size at the time of the visit.
   * Antidiabetic pharmacological treatment that patients currently take through the computer clinical history.
   * Changes in the antidiabetic pharmacological treatment, in the diet, in physical exercise and in sleep hygiene through a clinical interview with the patient.

   The instrument used is the PSQI that is a validated version in Spanish facilitated by its authors from the University of Pittsburgh. It consists of 24 items, 19 are answered by the patient and 5 are answered by the couple or roommate. In the event that the patient only goes to the consultation, only the first 19 items will be answered.

   The maximum score of the questionnaire is 21 points. Scores greater than five points indicate poor quality in the sleep standard.

   The questionnaires will be completed by the nursing professionals assigned to the patients through an individual, directed and structured interview, after explaining the study and justifying the access and review of the clinical history. The data collection will be by manual registration in a grill.

   The data collection will be made in the Primary Care Nursing consultation when the patient goes to a visit.

   The principal investigator will be responsible for the review of clinical histories to obtain the variables and analysis of the PSQI, noting the result in the clinical history.

   Two sections will be used in the registry of the information collected in the consultation to which the principal investigator has access.
   * General data section where all the variables mentioned above will be included.
   * Specific data section for PSQI analysis, in which the responses of the questionnaire will be introduced to obtain the variables of declared hours, sleep efficiency and the result.

   A screening visit and three follow-up visits will be carried out to each patient included in the study in which the professionals will follow a support guide by presenting the project to the team.
   * Screening visit:

     * Identify the patient with diagnosis prediabetes or DM2. Analyze inclusion and exclusion criteria.
     * Once included, explain the study and give a fact sheet.
     * Provide informed consent to be signed by the patient.
     * Pass the first PSQI. Patients with good sleep quality will be excluded.
     * Ask for previous HbA1c if the last one registered exceeds 6 months.
     * Schedule the patient in a month. The principal investigator will write down the result of the PSQI and the clinical order to follow
   * First visit:

     • Look at clinical course. The PSQI result and the clinical order will appear depending on the group to which the patient belongs (experimental or control).

     - Experimental: the educational intervention will be carried out and the booklet of Recommendations on Sleep Hygiene will be delivered.

     - Control: no educational intervention will be carried out.

     • Ask for the analysis of HbA1c and basal glycaemia to be done in the 3 months after in both groups.

     • Schedule the patient for results (3 months).
     * Schedule a telephone contact (1 month)
   * Second visit:

     * Carry out telephone contact as an educational reinforcement on sleep hygiene recommendations one month after the intervention.
   * Third visit:

     • Look at analytical results.
     * Ask about changes in the antidiabetic pharmacological treatment, diet, physical exercise and sleep hygiene.
     * Re-pass PSQI. The principal researcher will review the clinical history to obtain the variables to study. When the study ends at the last visit, the results of the PSQI will be re-analysed, as well as the remaining variables to perform the statistical analysis of the results and the final report of the study.

   First, the initial comparability of the groups will be checked by calculating the Student's T value and its statistical significance for the quantitative variables: basal glycemia, HbA1c, declared sleep hours, sleep efficiency, age and BMI. The variables: sex, diagnosis, PSQI and antidiabetic treatment will be compared by the significance of the chi-square test.

   The premise of randomness will remain intact, and patients will be analysed according to intention to treat.

   On the other hand, subsets of the study groups will be analysed (by sex, age group, treatment, BMI).

   As a global result of the clinical trial, the difference between the glycemia and HbA1c values of the final figure with respect to the initial one will be calculated with its respective 95% confidence interval within the intervention group and within the control group and the control group with respect to the group intervention, also with the 95% confidence interval.

   Through our study we want to corroborate the available evidence on the influence of sleep duration and quality on the ethology of DM2.

   There have been few studies in the field of Primary Care on the importance of sleep on the health of people. Sleeping is a health habit and, as such, is a tributary of educational interventions in the health environment.

   The scientific demonstration that a concrete measure of health education such as the one proposed in this study, is useful in demonstrable biological terms, would open a door to healthy sleep promotion activities in routine clinical practice.

   Regarding the socioeconomic aspect, information as a basis for health education and, specifically, in the topic of sleep hygiene does not require expensive resources and, through our study, we intend to demonstrate that it can be done from the primary care nursing consultation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Hb1Ac greater than or equal to 5.7% at the time of diagnosis.
* PSQI greater than 5 points (poor sleep quality).
* Acceptance of participation in the study.

Exclusion Criteria:

* People diagnosed with:

  * Obstructive Sleep Apnea Syndrome.
  * Narcolepsy
  * Fibromyalgia
  * Dementias
  * Schizophrenia
  * Psychosis
  * Major depression
* People with shift working hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change of glycated hemoglobin levels. | Three months
  Change the level of HbA1c in patients diagnosed with DM2 or prediabetes by an intervention in sleep hygiene.
  The levels will be measured by blood test according to laboratory protocol.

SECONDARY OUTCOMES:
Change in sleep quality: Pittsburgh Sleep Quality Index | Three months.
  Sleep quality will be measured with the Pittsburgh Sleep Quality Index before and after the intervention. The score varies between 0 and 21 points. A higher score means a worse quality of sleep. A total score less or equal than to five indicates that the quality of sleep is optimal, while a total score greater than five suggests that you have sleep problems.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina García Serrano, Nurse, Principal Investigator — Institut Català de la Salut; Jesús Pujol Salud, Doctor, Principal Investigator — Institut Català de la Salut; Lídia Aran Solé, Nurse, Principal Investigator — Institut Català de la Salut; Joaquim Sol, MSc, Principal Investigator — Institut Català de la Salut-IDIAP Jordi Gol
Locations (1):
- Centro Atención Primaria - Institut Català de la Salut, Balaguer, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed, the study protocol and results will be published in a scientific journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: The IPD sharing would require presentation of a study protocol in order to prove the consutant investigators work in the same research area.

REFERENCES:
- [Result] Chaput JP, Despres JP, Bouchard C, Tremblay A. Association of sleep duration with type 2 diabetes and impaired glucose tolerance. Diabetologia. 2007 Nov;50(11):2298-304. doi: 10.1007/s00125-007-0786-x. Epub 2007 Aug 24. PMID 17717644
- [Result] Morselli LL, Guyon A, Spiegel K. Sleep and metabolic function. Pflugers Arch. 2012 Jan;463(1):139-60. doi: 10.1007/s00424-011-1053-z. Epub 2011 Nov 19. PMID 22101912
- [Result] Ayas NT, White DP, Al-Delaimy WK, Manson JE, Stampfer MJ, Speizer FE, Patel S, Hu FB. A prospective study of self-reported sleep duration and incident diabetes in women. Diabetes Care. 2003 Feb;26(2):380-4. doi: 10.2337/diacare.26.2.380. PMID 12547866
- [Result] Tasali E, Leproult R, Ehrmann DA, Van Cauter E. Slow-wave sleep and the risk of type 2 diabetes in humans. Proc Natl Acad Sci U S A. 2008 Jan 22;105(3):1044-9. doi: 10.1073/pnas.0706446105. Epub 2008 Jan 2. PMID 18172212
- [Result] Yaggi HK, Araujo AB, McKinlay JB. Sleep duration as a risk factor for the development of type 2 diabetes. Diabetes Care. 2006 Mar;29(3):657-61. doi: 10.2337/diacare.29.03.06.dc05-0879. PMID 16505522
- [Result] Gottlieb DJ, Punjabi NM, Newman AB, Resnick HE, Redline S, Baldwin CM, Nieto FJ. Association of sleep time with diabetes mellitus and impaired glucose tolerance. Arch Intern Med. 2005 Apr 25;165(8):863-7. doi: 10.1001/archinte.165.8.863. PMID 15851636
- [Result] Gangwisch JE, Heymsfield SB, Boden-Albala B, Buijs RM, Kreier F, Pickering TG, Rundle AG, Zammit GK, Malaspina D. Sleep duration as a risk factor for diabetes incidence in a large U.S. sample. Sleep. 2007 Dec;30(12):1667-73. doi: 10.1093/sleep/30.12.1667. PMID 18246976
- [Result] Knutson KL, Ryden AM, Mander BA, Van Cauter E. Role of sleep duration and quality in the risk and severity of type 2 diabetes mellitus. Arch Intern Med. 2006 Sep 18;166(16):1768-74. doi: 10.1001/archinte.166.16.1768. PMID 16983057
- [Result] Mallon L, Broman JE, Hetta J. High incidence of diabetes in men with sleep complaints or short sleep duration: a 12-year follow-up study of a middle-aged population. Diabetes Care. 2005 Nov;28(11):2762-7. doi: 10.2337/diacare.28.11.2762. PMID 16249553
- [Result] Bjorkelund C, Bondyr-Carlsson D, Lapidus L, Lissner L, Mansson J, Skoog I, Bengtsson C. Sleep disturbances in midlife unrelated to 32-year diabetes incidence: the prospective population study of women in Gothenburg. Diabetes Care. 2005 Nov;28(11):2739-44. doi: 10.2337/diacare.28.11.2739. PMID 16249549
- [Result] Copinschi G, Leproult R, Spiegel K. The important role of sleep in metabolism. Front Horm Res. 2014;42:59-72. doi: 10.1159/000358858. Epub 2014 Apr 7. PMID 24732925
- [Result] Nedeltcheva AV, Scheer FA. Metabolic effects of sleep disruption, links to obesity and diabetes. Curr Opin Endocrinol Diabetes Obes. 2014 Aug;21(4):293-8. doi: 10.1097/MED.0000000000000082. PMID 24937041
- [Result] Stamatakis KA, Punjabi NM. Effects of sleep fragmentation on glucose metabolism in normal subjects. Chest. 2010 Jan;137(1):95-101. doi: 10.1378/chest.09-0791. Epub 2009 Jun 19. PMID 19542260
- [Result] Itani O, Jike M, Watanabe N, Kaneita Y. Short sleep duration and health outcomes: a systematic review, meta-analysis, and meta-regression. Sleep Med. 2017 Apr;32:246-256. doi: 10.1016/j.sleep.2016.08.006. Epub 2016 Aug 26. PMID 27743803
- [Result] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- See also: Ezkurra P. Guía de actualización en diabetes mellitus tipo 2. Fundación redGDPS. 2016. — http://redgdps.org/gestor/upload/GUIA2016/Guia_Actualizacion_2016.pdf
- See also: Instituto del Sueño. ¿Qué es el sueño? — http://www.iis.es/que-es-como-se-produce-el-sueno-fases-cuantas-horas-dormir/
- See also: Cunha MC, Zanetti ML, Hass VJ. Calidad del sueño en diabéticos tipo 2. Rev. Latino-Am. Enfermagem. 2008;16 (5): 850-855. — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0104-11692008000500009&lan=pt.g
- See also: SES. Pautas de actuación y seguimiento del Insomnio. 2016. — http://www.ses.org.es/docs/guia-de-insomnio-2016.pdf
- See also: Imazu MF, Nascimento B, Oliveira G, Aparecida C, Silva S. Efectividad de las intervenciones individual y en grupo en personas con diabetes tipo 2. Revista Latino-Americana de Enfermagem; 2015. 23(2) — http://www.scielo.br/pdf/rlae/v23n2/es_0104-1169-rlae-23-02-00200.pdf
- See also: Menor Rodríguez María, Aguilar Cordero María, Mur Villar Norma, Santana Mur Cinthya. Efectividad de las intervenciones educativas para la atención de la salud. Revisión sistemática. Medisur. 2017;15 (1):75-84. — http://scielo.sld.cu/scielo.php?script=sci_arttext&pid=S1727-897X2017000100011&lng=es.